CLINICAL TRIAL: NCT05479383
Title: Tobacco Use and Uptake of COVID-19 Vaccinations in Finland: a General Population Study
Brief Title: Tobacco Use and Uptake of COVID-19 Vaccinations
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Karolinska Institutet (Other); Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: THL/713/6.00.00/2021.2
Record Dates: First submitted 2022-07-28; First posted 2022-07-29 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; Smoking; Tobacco Use; Vaccination Refusal
Keywords: Tobacco use; Smoking; COVID-19; SARS-CoV-2; Vaccinations; Cohort studies
MeSH Terms: conditions — COVID-19; Smoking; Tobacco Use; Vaccination Refusal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tobacco users: Tobacco users
  Never smokers (reference group) will be compared with former smokers, occasional smokers and daily smokers.
  Never snus users (reference group) will also compare with never users, former users and current users.
  Interventions: Other: Not applicable, this is an observational study

INTERVENTIONS:
Other: Not applicable, this is an observational study — Not applicable, this is an observational study

SUMMARY:
This is an observational study of participants in two general population health surveys (FinSote 2018 and 2020) who are followed up for their COVID-19 vaccinations or end of follow-up. The primary objective is to examine the association between tobacco use and COVID-19 vaccine uptake and between-dose spacing.

DETAILED DESCRIPTION:
Most high income countries have rolled out COVID-19 vaccinations, with the promise of reducing incident COVID-19 infections and preventing hospitalizations and deaths. A high vaccination coverage is crucial for several reasons: (i) to reduce the number of new COVID-19 cases, (ii) to diminish selective pressures leading to the emergence of new variants of concern, (iii) to prevent severe COVID-19 outcomes, such as hospitalizations and deaths, and (iv) to potentially reduce the risk of post-acute COVID-19 symptoms.

Smokers are at higher risk of COVID-19 hospitalizations and deaths and might thus benefit greatly from high vaccination coverage. However, evidence suggests that they may be less likely to be vaccinated, as smokers are less likely to adhere to preventive measures in general and have lower adherence to other vaccines. Reports of a protective role of smoking on the risk of COVID-19 infection might have also reduced the perceived risks from being infected.

Evidence regarding tobacco use and COVID-19 vaccine hesitancy is mixed. Some studies have shown greater mistrust in COVID-19 vaccine benefits and greater vaccine hesitancy and lower vaccine acceptance compared to non-smokers, while other studies have reported no differences by smoking status or lower levels of vaccine hesitancy in smokers compared to non-smokers. Few studies have examined the relationship between tobacco use and vaccine uptake, showing that smokers had higher odds of being vaccinated. These studies, however, are not representative of the general population and relied on self-reported vaccination status, resulting in higher risk of selection and information bias.

The investigators will expand current knowledge by examining two forms of tobacco use in Finland -smoking and smokeless tobacco use (snus)- and by analysing the spacing between vaccine doses. The study will use data from nationally representative surveys in Finland linked to vaccination registries, which reduces the risk of selection and information bias.

ELIGIBILITY:
Inclusion Criteria:

* Permanent residents of Finland
* Registered in the Population Register at the moment of sampling
* Aged 20 and over
* Participated in the FinSote surveys in 2018 or 2020
* Provided consent for register linkage

Exclusion Criteria:

* Temporary residents in Finland or tourists
* Age less than 20 years old
* Did not participate in FinSote surveys in 2018, 2019 and 2020
* Did not provide consent for register linkage

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Permanent residents in Finland aged 20 and over who participated in the FinSote surveys in 2018 and 2020. These are general population samples representative of the Finnish population. The sampling frame was the Population Register (in 2020 the Digital and Population Data Services Agency, created after the merge between the Population Register of Statistics Finland and local register offices), which includes all individuals residing permanently in Finland, including conscripts and people living in institutions.
Sampling Method: Probability Sample
Enrollment: 42935 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Vaccination uptake of at least two doses of a COVID-19 vaccine | Baseline until date of vaccination or May 31, 2022
  Proportion of participants with at least two doses of a COVID-19 vaccine

SECONDARY OUTCOMES:
Vaccination uptake of at least one dose of a COVID-19 vaccine | Baseline until date of vaccination or May 31, 2022
  Proportion of participants with at least one dose of a COVID-19 vaccine
Vaccination uptake of complete COVID-19 vaccination scheme (two doses and a booster dose) | Baseline until date of vaccination or May 31, 2022
  Proportion of participants with two doses and a booster dose of a COVID-19 vaccine
Spacing of first and second COVID-19 dose | Baseline until date of vaccination or May 31, 2022
  Proportion of participants with more than 7 months between the first and second COVID-19 dose
Spacing of second dose and booster dose of the COVID-19 vaccine | Baseline until date of vaccination or May 31, 2022
  Proportion of participants with more than 7 months between the second dose and booster dose of the COVID-19 vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Sakari Karvonen, PhD, Principal Investigator — Finnish Institute for Health and Welfare
Locations (1):
- Finnish Institute for Health and Welfare, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No
Researchers can access individual data by contacting the Responsible Researcher at the Finnish Institute for Health and Welfare, Suvi Parikka, suvi.parikka [at] thl.fi.
  Information about FinSote surveys, including questionnaires, can be found in https://thl.fi/fi/tutkimus-ja-kehittaminen/tutkimukset-ja-hankkeet/finsote-tutkimus

REFERENCES:
- [Background] Simons D, Shahab L, Brown J, Perski O. The association of smoking status with SARS-CoV-2 infection, hospitalization and mortality from COVID-19: a living rapid evidence review with Bayesian meta-analyses (version 7). Addiction. 2021 Jun;116(6):1319-1368. doi: 10.1111/add.15276. Epub 2020 Nov 17. PMID 33007104
- [Background] Jackson SE, Paul E, Brown J, Steptoe A, Fancourt D. Negative Vaccine Attitudes and Intentions to Vaccinate Against Covid-19 in Relation to Smoking Status: A Population Survey of UK Adults. Nicotine Tob Res. 2021 Aug 18;23(9):1623-1628. doi: 10.1093/ntr/ntab039. PMID 33751125
- [Background] Krebs NM, D'Souza G, Bordner C, Allen SI, Hobkirk AL, Foulds J, Yingst JM. COVID-19 Vaccination Uptake and Hesitancy Among Current Tobacco Users. Tob Use Insights. 2021 Dec 20;14:1179173X211068027. doi: 10.1177/1179173X211068027. eCollection 2021. PMID 34987300
- [Background] Ali M, Ahmed S, Bonna AS, Sarkar AS, Islam MA, Urmi TA, Proma TS. Parental coronavirus disease vaccine hesitancy for children in Bangladesh: a cross-sectional study. F1000Res. 2022 Jan 25;11:90. doi: 10.12688/f1000research.76181.2. eCollection 2022. PMID 35211297
- [Background] Oruc MA, Ozturk O. Attitudes of health care professionals towards COVID-19 vaccine - a sequence from Turkey. Hum Vaccin Immunother. 2021 Oct 3;17(10):3377-3383. doi: 10.1080/21645515.2021.1928462. Epub 2021 Jun 18. PMID 34142925
- [Background] Wu J, Li Q, Silver Tarimo C, Wang M, Gu J, Wei W, Ma M, Zhao L, Mu Z, Miao Y. COVID-19 Vaccine Hesitancy Among Chinese Population: A Large-Scale National Study. Front Immunol. 2021 Nov 29;12:781161. doi: 10.3389/fimmu.2021.781161. eCollection 2021. PMID 34912346
- [Background] Luk TT, Zhao S, Wu Y, Wong JY, Wang MP, Lam TH. Prevalence and determinants of SARS-CoV-2 vaccine hesitancy in Hong Kong: A population-based survey. Vaccine. 2021 Jun 16;39(27):3602-3607. doi: 10.1016/j.vaccine.2021.05.036. Epub 2021 May 18. PMID 34034950
- [Background] Wisniak A, Baysson H, Pullen N, Nehme M, Pennacchio F, Zaballa ME, Guessous I, Stringhini S; Specchio-COVID19 study group. COVID-19 vaccination acceptance in the canton of Geneva: a cross-sectional population-based study. Swiss Med Wkly. 2021 Dec 14;151:w30080. doi: 10.4414/smw.2021.w30080. eCollection 2021 Dec 6. PMID 34908389
- [Background] Ishimaru T, Okawara M, Ando H, Hino A, Nagata T, Tateishi S, Tsuji M, Matsuda S, Fujino Y; CORoNaWork Project. Gender differences in the determinants of willingness to get the COVID-19 vaccine among the working-age population in Japan. Hum Vaccin Immunother. 2021 Nov 2;17(11):3975-3981. doi: 10.1080/21645515.2021.1947098. Epub 2021 Jul 2. PMID 34213406
- [Background] Ko T, Dendle C, Woolley I, Morand E, Antony A. SARS-COV-2 vaccine acceptance in patients with rheumatic diseases: a cross-sectional study. Hum Vaccin Immunother. 2021 Nov 2;17(11):4048-4056. doi: 10.1080/21645515.2021.1958611. Epub 2021 Aug 6. PMID 34357827
- [Background] Tan LF, Huak CY, Siow I, Tan AJ, Venugopalan PM, Premkumar A, Seetharaman SK, Tan BYQ. The road to achieving herd immunity: factors associated with Singapore residents' uptake and hesitancy of the COVID-19 vaccination. Expert Rev Vaccines. 2022 Apr;21(4):561-567. doi: 10.1080/14760584.2022.2021883. Epub 2022 Jan 11. PMID 34937504
- [Background] Tiirinki H, Viita-Aho M, Tynkkynen LK, Sovala M, Jormanainen V, Keskimaki I. COVID-19 in Finland: Vaccination strategy as part of the wider governing of the pandemic. Health Policy Technol. 2022 Jun;11(2):100631. doi: 10.1016/j.hlpt.2022.100631. Epub 2022 Apr 14. PMID 35437478
- [Derived] Pena S, Zhou Z, Kestila L, Galanti MR, Shaaban AN, Caspersen IH, Magnus P, Geraldo P, Rojas-Saunero P, Parikka S, Nohynek H, Karvonen S. Tobacco Use and Uptake of COVID-19 Vaccinations in Finland: A Population-Based Study. Nicotine Tob Res. 2024 Oct 22;26(11):1553-1562. doi: 10.1093/ntr/ntad234. PMID 38196092
- See also: Description of the Tobrisk-CoV project — https://www.nordforsk.org/projects/addressing-smoking-paradox-etiology-covid-19-through-population-based-studies-tobrisk-cov

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT05479383/Prot_SAP_002.pdf